CLINICAL TRIAL: NCT02925585
Title: Vaginal Tactile Imaging in Assessment of Pelvic Floor Conditions
Brief Title: Vaginal Tactile Imaging for Pelvic Floor Prolapse
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: VTI09; SB1AG034714 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre/post pelvic floor surgery imaging
  Interventions: Other: Pre/post imaging

INTERVENTIONS:
Other: Pre/post imaging

SUMMARY:
The investigators will analyze biomechanical transformation of pelvic floor tissues and support structures under affected pelvic floor conditions and repaired states after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female of 21 years or older, and
2. No prior pelvic floor surgery, and
3. One of the following:

Normal pelvic floor conditions, or POP Stage I affecting one or more vaginal compartment, or POP Stage II affecting one or more vaginal compartment, or POP Stage III affecting one or more vaginal compartment, or POP Stage IV affecting one or more vaginal compartment

Exclusion Criteria:

1. Active skin infection or ulceration within the vagina
2. Presence of a vaginal septum;
3. Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder;
4. Ongoing radiation therapy for pelvic cancer;
5. Impacted stool;
6. Significant pre-existing pelvic pain including levator ani syndrome, severe vaginismus or vulvadynia;
7. Severe hemorrhoids;
8. Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician;
9. Current pregnancy.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for pelvic floor surgery
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Tissue elasticity change after the surgery measured as a gradient in tactile image. Unit of measure: mmHg/mm | pre-surgery and post-surgery (4-6 months after surgery) measurements
  Tissue elasticity is measured for entire anterior and posterior compartments
Pelvic floor muscle strength change after the surgery measured as a pressure dynamic feedback during muscle contractions. Unit of measure: mmHg | pre-surgery and post-surgery (4-6 months after surgery) measurements
  Muscle strength is measured during voluntary and involuntary muscle contractions, involuntary relaxation and Valsalva maneuver.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Pelvic Floor Institute, Tampa, Florida
  - Princeton Urogynecology PU, Princeton, New Jersey
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Inova Health System Foundation, Falls Church, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Scientific Publications of the study results